CLINICAL TRIAL: NCT06053541
Title: Hospitalization, Mortality Rates and Costs Associated With Chronic Obstructive Pulmonary Disease (COPD) in Distrito Federal, Brazil, Before and After the Change in 2018 State COPD Protocol Version - Real-world Data
Brief Title: Morbid Rates After Spiriva Chronic Obstructive Pulmonary Disease (COPD) Protocol Change
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0205-0548
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with COPD, admitted to the hospital with acute exacerbations: Patients over 40 years of age, diagnosed with Chronic Obstructive Pulmonary Disease (COPD), admitted to the hospital with acute exacerbations as recorded in the DATASUS (Unified Health Brazilian System Informatics Department (in Portuguese) between August 2017 and July 2019. Patients were treated with either Tiotropium bromide in soft mist inhaler (SPIRIVA® RESPIMAT®) or with Glycopyrronium bromide in dry powder inhaler (Seebri® Breezhaler®) as part of the treatment plan for Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Distrito Federal (DF) in Brazil.

SUMMARY:
This study evaluates hospitalizations and mortality in patients with Chronic Obstructive Pulmonary Disease (COPD) before and after the implantation of a new COPD treatment plan (replacement of tiotropium soft mist inhaler for glycopyrronium dry powder inhaler) by the Health State Secretariat of Federal District in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 40 years of age at the time of hospital admission
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) according to the International Statistical Classification of Diseases and Related Health Problems Version 10 (ICD-10) established by the Health Care Protocol of the Health Secretariat of Federal District (SES/DF), with the following codes:

  * J41.0 - Simple chronic bronchitis
  * J41.1 - Mucopurulent chronic bronchitis
  * J41.8 - Mixed simple and mucopurulent chronic bronchitis
  * J42 - Unspecified chronic bronchitis
  * J43.1 - Panlobular emphysema
  * J43.2 - Centrilobular emphysema
  * J43.8 - Other emphysema
  * J43.9 - Emphysema, unspecified
  * J44.0 - Chronic obstructive pulmonary disease with acute lower respiratory infection
  * J44.1 - Chronic obstructive pulmonary disease with acute exacerbation, unspecified
  * J44.8 - Other specified chronic obstructive pulmonary disease
  * J44.9 - Chronic obstructive pulmonary disease, unspecified

Exclusion Criteria:

* Patients younger than 40 yeas of age at the time of hospital admission

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 40 years of age, diagnosed with Chronic Obstructive Pulmonary Disease (COPD), admitted to the hospital with acute exacerbations of the disease between August 2017 and July 2019 in Federal District, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 3015000 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim Brasil, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study based on existing data from the Brazilian Public Healthcare System (SUS) to investigate the potential different patterns on chronic obstructive pulmonary disease (COPD) mortality, hospitalizations, ICU usage rates and costs after the COPD protocol change in Distrito Federal (DF), Brazil, in August 2018, with a substitution of tiotropium in soft mist inhaler to glycopyrronium in dry powder inhaler.
Pre-assignment Details: The SUS data was not individualized, this study had access to the total number of hospitalizations and not to the exact number of patients as the same patient could be hospitalized more than once a year.
Period: Overall Study
Arm/Group | Patients Diagnosed With COPD, Admitted to the Hospital With Acute Exacerbations
Started | 3015000
Completed | 3015000
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Distrito Federal (DF) in Brazil who were hospitalized between August 2017 and July 2019.
Units Other Than Participants: Hospitalizations
Arm/Group | Patients Diagnosed With COPD, Admitted to the Hospital With Acute Exacerbations
Number analyzed (Participants) | 3015000
Number analyzed (Hospitalizations) | 1430
Age, Customized [Count of Units; unit: Hospitalizations]
  40 to 59 years old | 198
  60 to 79 years old | 876
  Over 80 years old | 876
Sex: Female, Male [Count of Units; unit: Hospitalizations] — Sex is reported per patient hospitalization entry Population: Sex is reported per patient hospitalization entry, as the SUS data was not individualized, this study had access to the total number of hospitalizations and not to the exact number of patients, the same patient could be hospitalized more than once a year.
  Hospitalizations
    number analyzed (Participants) | 1430
    Female | 741
    Male | 689
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Hospital Admissions in Chronic Obstructive Pulmonary Disease (COPD) Patients
Description: Number of hospital admissions in Chronic Obstructive Pulmonary Disease (COPD) patients, is reported, the same patient could be hospitalized more than once a year.
Time Frame: From August 2017 to July 2018 (Tiotropium treatment - MAT1 period) and August 2018 to July 2019 (Glycopyrronium treatment - MAT2 Period), Up to 1 year.
Population: Patients with Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Federal District in Brazil who were hospitalized between August 2017 and July 2019. Federal District 2019 population was 3015000 according to the Brazilian Institute of Geography and Statistics.
Measure: Number; unit: Hospitalizations
Units Other Than Participants: Hospitalizations
Groups:
- Tiotropium Treatment - MAT1: In the MAT1 (total arithmetic mean 1) period, August 2017 to July 2018 data cut available in the DATASUS (Unified Health Brazilian System Informatics Department (in Portuguese)) hospitalizations, patients received Tiotropium bromide in soft mist inhaler (SPIRIVA® RESPIMAT®) as part of the treatment plan for Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Distrito Federal (DF) in Brazil.
- Glycopyrronium Treatment - MAT2: In the MAT2 (total arithmetic mean 2) period, August 2018 to July 2019 data cut available in the DATASUS (Unified Health Brazilian System Informatics Department (in Portuguese) hospitalizations, patients received Glycopyrronium bromide in dry powder inhaler (Seebri® Breezhaler®) as part of the treatment plan for Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Distrito Federal (DF) in Brazil.
Arm/Group | Tiotropium Treatment - MAT1 | Glycopyrronium Treatment - MAT2
Number analyzed (Participants) | 3015000 | 3015000
Number analyzed (Hospitalizations) | 665 | 765
Hospitalizations | 665 | 765
Statistical Analysis 1: Comparison: Tiotropium Treatment - MAT1 vs Glycopyrronium Treatment - MAT2; For the evaluation of statistical significance, considering that the data do not follow a normal distribution and that the two samples are independent and not paired, the Mann-Whitney test was applied and a p value < 0.05 was considered; Test type: Other; p = 0.24, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Deaths of Hospitalized Chronic Obstructive Pulmonary Disease (COPD) Patients
Description: Number of deaths of hospitalized Chronic Obstructive Pulmonary Disease (COPD) patients, the same patient could be hospitalized more than once a year.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Deaths
Units Other Than Participants: Hospitalizations
Groups:
- Tiotropium Treatment - MAT1: In the MAT1 (total arithmetic mean 1) period, August 2017 to July 2018 data cut available in the DATASUS (Unified Health Brazilian System Informatics Department (in Portuguese)), patients received Tiotropium bromide in soft mist inhaler (SPIRIVA® RESPIMAT®) as part of the treatment plan for Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Distrito Federal (DF) in Brazil.
- Glycopyrronium Treatment - MAT2: In the MAT2 (total arithmetic mean 2) period, August 2018 to July 2019 data cut available in the DATASUS (Unified Health Brazilian System Informatics Department (in Portuguese), patients received Glycopyrronium bromide in dry powder inhaler (Seebri® Breezhaler®) as part of the treatment plan for Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Distrito Federal (DF) in Brazil.
Arm/Group | Tiotropium Treatment - MAT1 | Glycopyrronium Treatment - MAT2
Number analyzed (Participants) | 3015000 | 3015000
Number analyzed (Hospitalizations) | 665 | 765
Deaths | 52 | 67
Statistical Analysis 1: Comparison: Tiotropium Treatment - MAT1 vs Glycopyrronium Treatment - MAT2; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.37, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Total Costs Associated With Chronic Obstructive Pulmonary Disease (COPD) Hospitalizations
Description: Total accumulated costs to the payer per year associated with Chronic Obstructive Pulmonary Disease (COPD) hospitalizations, is reported, the same patient could have been hospitalized more than once a year. No individual costs, the cost reported are the total spent per year.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Brazilian Reais (R$)
Units Other Than Participants: Hospitalizations
Arm/Group | Tiotropium Treatment - MAT1 | Glycopyrronium Treatment - MAT2
Number analyzed (Participants) | 3015000 | 3015000
Number analyzed (Hospitalizations) | 665 | 765
Brazilian Reais (R$) | 828761.94 | 1267318.42
Statistical Analysis 1: Comparison: Tiotropium Treatment - MAT1 vs Glycopyrronium Treatment - MAT2; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Infirmary Beds
Description: Average monthly number of available Infirmary beds, including available general and ICU (Intensive care unit) beds are reported, the same patient could have been hospitalized more than once a year.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beds
Units Other Than Participants: Hospitalizations
Arm/Group | Tiotropium Treatment - MAT1 | Glycopyrronium Treatment - MAT2
Number analyzed (Participants) | 3015000 | 3015000
Number analyzed (Hospitalizations) | 665 | 765
Beds
  Beds in the general practice and Pulmonology: number analyzed (Hospitalizations) | 665 | 465
  Beds in the general practice and Pulmonology | 883.8 (21.2) | 895.5 (17.7)
  Beds in Adults ICU: number analyzed (Hospitalizations) | 665 | 665
  Beds in Adults ICU | 150.7 (1.2) | 146.6 (1.0)
Statistical Analysis 1: Comparison: Tiotropium Treatment - MAT1 vs Glycopyrronium Treatment - MAT2; Beds in the general practice and Pulmonology: For the evaluation of statistical significance, considering that the data do not follow a normal distribution and that the two samples are independent and not paired, the Mann-Whitney test was applied and a p value < 0.05 was considered; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tiotropium Treatment - MAT1 vs Glycopyrronium Treatment - MAT2; Beds in Adults ICU: For the evaluation of statistical significance, considering that the data do not follow a normal distribution and that the two samples are independent and not paired, the Mann-Whitney test was applied and a p value < 0.05 was considered; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Hospitalizations With Intensive Care Unit (ICU) Admissions Over Total Number of Hospitalizations
Description: Number of hospitalizations with intensive care unit (ICU) admissions over total number of hospitalizations, is reported, the same patient could have been hospitalized more than once a year.
Time Frame: as for outcome 1
Population: Patients with Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Distrito Federal (DF) in Brazil who were hospitalized between August 2017 and July 2019. The Federal District 2019 population was 3015000 according to the Brazilian Institute of Geography and Statistics.
Measure: Number; unit: Hospitalizations
Units Other Than Participants: Hospitalization entries
Arm/Group | Tiotropium Treatment - MAT1 | Glycopyrronium Treatment - MAT2
Number analyzed (Participants) | 3015000 | 3015000
Number analyzed (Hospitalization entries) | 665 | 765
Hospitalizations | 16 | 37
Statistical Analysis 1: Comparison: Tiotropium Treatment - MAT1 vs Glycopyrronium Treatment - MAT2; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Total Costs Associated With Chronic Obstructive Pulmonary Disease (COPD) Hospitalizations With Admission to Intensive Care Unit (ICU)
Description: Total costs associated with Chronic Obstructive Pulmonary Disease (COPD) hospitalizations with admission to intensive care unit (ICU) , is reported, the same patient could have been hospitalized more than once a year.
Time Frame: as for outcome 1
Population: Patients with Chronic Obstructive Pulmonary Disease (COPD) defined by the Health State Secretariat of Distrito Federal (DF) in Brazil who were hospitalized between August 2017 and July 2019. Patient hospitalizations with intensive care unit (ICU) admissions were analyzed. The Federal District 2019 population was 3015000 according to the Brazilian Institute of Geography and Statistics.
Measure: Number; unit: Brazilian Reais (R$)
Units Other Than Participants: Hospitalization with ICU admissions
Arm/Group | Tiotropium Treatment - MAT1 | Glycopyrronium Treatment - MAT2
Number analyzed (Participants) | 3015000 | 3015000
Number analyzed (Hospitalization with ICU admissions) | 16 | 37
Brazilian Reais (R$) | 149145.17 | 298051.06
Statistical Analysis 1: Comparison: Tiotropium Treatment - MAT1 vs Glycopyrronium Treatment - MAT2; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.07, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Not applicable for other Adverse Events (AEs) and serious AEs. All-Cause mortality was recorded for any hospitalization between August 2017 and July 2019, up to 2 years.
Description: This is a study with secondary use of data, safety reporting on an individual case level is not applicable. This study had access to the number of hospitalizations and not to the exact number of patients. Other Adverse Events (AEs) and Serious AEs were not collected. "0" total Number of Participants at Risk means not collected. All-cause mortality was reported based on the number of hospitalizations, the corresponding number at risk indicates the total number of hospitalizations recorded.
Arm/Group | Tiotropium Treatment - MAT1 | Glycopyrronium Treatment - MAT2
All-Cause Mortality (participants affected / at risk) | 52/665 | 67/765
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT06053541/Prot_SAP_000.pdf